CLINICAL TRIAL: NCT02731976
Title: The Influence of a Short-term Gluten-free Diet on the Human Gut Microbiome
Brief Title: Microbiome Composition Changes on 4 Week Gluten-free Diet Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M12.113965
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Human Microbiome
Keywords: Gluten-Free diet; Healthy individuals
MeSH Terms: interventions — Diet Therapy

ARMS (1):
- GFD (Experimental): After instruction of a dietician, participants adhered to a gluten-free diet for 4 weeks.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention

SUMMARY:
Changes in the gut microbiomes of healthy volunteers who followed a gluten-free diet (GFD) for four weeks were studied. Per participant, nine stool samples were collected: one at baseline, four during the GFD period, and four when they returned to their habitual diet. Microbiome profiles were determined using 16S rRNA sequencing and the samples were next processed for taxonomic and imputed functional composition. Additionally, participants kept a 3-day food diary and six gut health-related biomarkers were measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants aged >=16

Exclusion Criteria:

* Known gastrointestinal disorder
* Known food intolerance

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition upon gluten-free diet intervention | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet

SECONDARY OUTCOMES:
Changes in gut associated biomarker levels: fecal calprotectin | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: IL-1beta | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal human beta defensin 2 | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal chromogranin A | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal short chain fatty acids: propionate | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma citrulline | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal short chain fatty acids: acetate | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal short chain fatty acids: butyrate | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal short chain fatty acids: valerate | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: fecal short chain fatty acids: caproate | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: IL-6 | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: IL-8 | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: IL-10 | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: IL-12 | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet
Changes in gut associated biomarker levels: plasma cytokines: TNFalpha | baseline, 4 weeks gluten-free diet and 4 weeks habitual diet

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Result] Baranska A, Tigchelaar E, Smolinska A, Dallinga JW, Moonen EJ, Dekens JA, Wijmenga C, Zhernakova A, van Schooten FJ. Profile of volatile organic compounds in exhaled breath changes as a result of gluten-free diet. J Breath Res. 2013 Sep;7(3):037104. doi: 10.1088/1752-7155/7/3/037104. Epub 2013 Jun 18. PMID 23774130